CLINICAL TRIAL: NCT02366546
Title: Multi-center, Investigator Initiated Phase 1 Study of NY-ESO-1 Specific TCR Gene Transferred T Lymphocytes With Solid Tumors
Brief Title: Investigator Initiated Phase 1 Study of TBI-1301
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mie University (Other)
Collaborators: Takara Bio Inc. (Industry); Shionogi (Industry); Fiverings Co., Ltd. (Other); Statcom Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Shinichi Kageyama, Professor, Mie University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1301-01
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumors
Keywords: Adoptive cell transfer; Cell therapy; Immunotherapy; NY-ESO-1; Esophageal cancer; Melanoma; Head and neck cancer; Ovarian cancer; Synovial sarcoma; TCR gene therapy
MeSH Terms: conditions — Esophageal Neoplasms; Melanoma; Head and Neck Neoplasms; Ovarian Neoplasms; Sarcoma, Synovial | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose TBI-1301 with pre-treatment 1 (Experimental): TBI-1301(5*10^8) single-dose administration with pre-treatment of cyclophosphamide alone.
  Interventions: Drug: TBI-1301; Drug: Cyclophosphamide
- High dose TBI-1301 with pre-treatment 1 (Experimental): TBI-1301(5*10^9) single-dose administration with pre-treatment of cyclophosphamide alone.
  Interventions: Drug: TBI-1301; Drug: Cyclophosphamide
- High dose TBI-1301 with pre-treatment 2 (Experimental): TBI-1301(5*10^9) single-dose administration with pre-treatment of cyclophosphamide and fludarabine.
  Interventions: Drug: TBI-1301; Drug: Cyclophosphamide; Drug: Fludarabine
- TBI-1301 with pre-treatment 1 or 2 (Experimental): Arm1, 2 or 3, which is considered as optimal.
  Interventions: Drug: TBI-1301; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: TBI-1301 — TBI-1301(5*10^8 or 5*10^9) is administered.
  Other Names: NY-ESO-1-specific TCR gene transduced T lymphocytes
Drug: Cyclophosphamide — Cyclophosphamide (750mg/m2/day x 2 days Intravenous (IV)) is administered as pre-treatment medication of TBI-1301.
  Other Names: Endoxan
Drug: Fludarabine — Fludarabine (20mg/m2 x 5 days Intravenous(IV)) is administered as pre-treatment medication of TBI-1301 in combination with cyclophosphamide.
  Other Names: Fludara
  Arms: High dose TBI-1301 with pre-treatment 2; TBI-1301 with pre-treatment 1 or 2

SUMMARY:
Following pre-treatment with cyclophosphamide and/or fludarabine, NY-ESO-1-specific TCR gene transduced T lymphocytes are transferred to the patients with NY-ESO-1-expressing solid tumors.

DETAILED DESCRIPTION:
Following pre-treatment with cyclophosphamide alone or in combination with fludarabine, NY-ESO-1-specific TCR gene transduced T lymphocytes are transferred to HLA-A*02:01 or HLA-A*02:06 positive patients with solid tumors which are 1) unresectable, refractory to standard therapy (chemotherapy, radiotherapy, etc), and 2) NY-ESO-1-expressing. The primary objective is to evaluate the safety and in vivo kinetics, and the secondary is to evaluate clinical effect.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumors
2. Solid tumor, which is unresectable, refractory to standard therapy (chemotherapy, radiotherapy, etc)
3. HLA-A*02:01 or HLA-A*02:06 positive
4. NY-ESO-1-expression by PCR or immunohistochemistry
5. ECOG Performance Status, 0 or 1
6. Age >=20 years on consent
7. No treatment (surgery, chemotherapy, radiotherapy, etc.) and expected sufficient recovery from the treatment at the time of the lymphocytes collection for gene transfer.
8. Life expectancy >=16 weeks after consent
9. No severe damage on the major organs (bone marrow, heart, lung, liver, kidney, etc) and meet the following lab value criteria:

   * WBC >= 2,500/μL
   * Hemoglobin >= 8.0g/dL
   * Platelets >= 75,000/μL
   * T. bilirubin < 1.5 x ULN
   * AST(GOT), ALT(GPT) < 3.0 x ULN
   * Creatinine < 1.5 x ULN
10. Ability to understand the study contents and to give a written consent at his/her free will.

Exclusion Criteria:

1. The following serious complications are excluded from the study;

   * Unstable angina, cardiac infarction, or heart failure
   * Uncontrolled diabetes or hypertension
   * Active infection
   * Obvious interstitial pneumonia or lung fibrosis by chest X-ray
   * Active autoimmune disease requiring steroids or immunosuppressive therapy.
2. Serious hypersensitivity
3. Tumor cell invasion into CNS
4. Active multiple cancer
5. Positive for HBs antigen or HBV-DNA observed in serum
6. Positive for HCV antibody and HCV-RNA observed in serum
7. Positive for antibodies against HIV or HTLV-1
8. Left Ventricular Ejection Fraction (LVEF): <= 50％
9. Percutaneous Oxygen saturation: < 94％
10. History of serious hypersensitivity reactions to bovine or murine derived substances.
11. History of hypersensitivity reaction to drugs used in this study.
12. Psychological disorder or drug dependency which may have impact on the consent.
13. Pregnant females, lactating females (except when they cease and don't resume lactation) or female and male patients who cannot agree to practice the adequate birth control after the consent during the study
14. Clinically significant systemic illness that in the judgment of the PI or sub-investigator would compromise the patient's ability to tolerate protocol therapy or significantly increase the risk of complications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Incidence and grade of adverse events (CTCAE) | 4 weeks
  • Confirm the toxicity profile, which is measured by the degree of grade and seriousness, duration, causality, classification, etc. of the adverse events.
Appearance of replication competent retrovirus by PCR | 4 weeks
  Confirm no replication competent retrovirus observed.
Appearance of clonality by LAM-PCR | 4 weeks
  Confirm no clonality is observed.
Kinetics of TBI-1301 in blood by realtime-PCR | 8 weeks
  Evaluate persistence and expansion of transferred TBI-1301.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Shiku, M.D., Ph.D., Study Chair — Department of Immuno-Gene Therapy, Mie University, Graduate School of Medicine Mie University Hospital; Shinichi Kageyama, M.D., Ph.D., Principal Investigator — Department of Immuno-Gene Therapy, Mie University, Graduate School of Medicine Mie University Hospital
Locations (1):
- Mie University Hospital, Tsu, Mie-ken, Japan

REFERENCES:
- [Derived] Ishihara M, Kitano S, Kageyama S, Miyahara Y, Yamamoto N, Kato H, Mishima H, Hattori H, Funakoshi T, Kojima T, Sasada T, Sato E, Okamoto S, Tomura D, Nukaya I, Chono H, Mineno J, Kairi MF, Diem Hoang Nguyen P, Simoni Y, Nardin A, Newell E, Fehlings M, Ikeda H, Watanabe T, Shiku H. NY-ESO-1-specific redirected T cells with endogenous TCR knockdown mediate tumor response and cytokine release syndrome. J Immunother Cancer. 2022 Jun;10(6):e003811. doi: 10.1136/jitc-2021-003811. PMID 35768164